CLINICAL TRIAL: NCT02675660
Title: Study to Evaluate the Safety, Tolerability, Kinetics, and Dynamics of Single and Multiple Doses of an Oral Formulation of L-Homoarginine
Brief Title: Single and Multiple Doses of an Oral Formulation of L-Homoarginine in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Homoarginine-UKE-KP2012-01
Record Dates: First submitted 2016-01-13; First posted 2016-02-05 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: kinetic data; volunteers
MeSH Terms: interventions — omega-N-aminohomoarginine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-Homoarginine (Experimental): 125 mg of L-homoarginine
  Interventions: Dietary Supplement: L-Homoarginine
- Placebo (Placebo Comparator): placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: L-Homoarginine — 125 mg L-homoarginine once daily
  Arms: L-Homoarginine
Drug: Placebo — placebo capsules once daily
  Arms: Placebo

SUMMARY:
This study represents an initial clinical evaluation of an oral formulation of L-homoarginine. L-homoarginine and L-arginine are amino acids found in food proteins and are both substrates for nitric oxide synthase (NOS). L-arginine is available as over the counter nutraceutical. This study will provide information on the dosing of L-homoarginine in order to reach high physiological plasma concentrations in humans.

DETAILED DESCRIPTION:
1. Study Design In a randomized, double-blind, placebo-controlled cross-over design participants receive either L-homoarginine 125 mg or placebo once daily in the morning for four weeks each. The study periods are separated by a washout phase of four weeks, and the sequence of the medications is randomly chosen in each participant. The study is preceded by a run-in phase, where all participant receive a single dose of 125 mg L-homoarginine. Blood samples (2.7 ml ethylenediaminetetraacetic acid vacutainer) for plasma L-homoarginine determinations are drawn at time points 0, 15 min, 30 min, 1, 2, 4, 8, 24, 48, 72, and 120 hours after single and multiple doses of L-homoarginine and placebo, respectively. At baseline and four weeks after each supplementation period (hArg and placebo), routine laboratory, arginine, asymmetric dimethylarginine, pulse wave velocity, augmentation index, flow-mediated vasodilatation, transcranial magnetic stimulation, and test battery of attentional performance are evaluated as secondary endpoints.
2. Study Duration One year
3. Sample Size Calculation and Statistical Evaluation Due to the exploratory nature of this pilot study, exploratory statistical methods will be used for statistical evaluation of the study results, and no formal sample size calculation was performed. In a previous study 20 participants were included to assess the kinetic, dynamic, and safety profile of L-citrulline and L-arginine [Schwedhelm et al. 2007]. Statistical comparisons will be performed using two-sided tests, i.e. Student's t-test and ANOVA. A p < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 20-75 years of age on the day of dosing and is generally healthy as determined by medical history, physical examination, and laboratory test values
2. For females, postmenopausal for at least 2 years prior to screening (confirmed by a negative hormone panel, i.e., plasma 17β-estradiol concentration of <20 pg/mL and follicle-stimulating hormone level of >40 IU/mL) or contraception
3. Has signed and received a copy of the written informed consent form approved by the investigator's Independent Ethics Committee (IEC), understands the purposes and risks of the study and agrees to follow the restrictions and schedule of procedures as defined by the study protocol

Exclusion Criteria:

1. Sitting blood pressure greater than 160/100 or less than 90/60 mm Hg
2. Sitting heart rate greater than 99 bpm or less than 50 beats per minute (bpm)
3. History of clinically significant hypotensive episodes or symptoms of fainting, dizziness, or light-headedness
4. Body Mass Index (BMI) greater than 32 or less than 16 at screening [BMI = Weight (kg) ÷ Height2 (m2)]
5. History or symptoms of cardiovascular disease, particularly coronary artery disease, arrhythmias,or congestive heart failure
6. History of significant central nervous system disease, including transient ischemic attack, stroke, seizure disorder, or behavioral disturbances

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 1 Month
  To determine the AUC of L-homoarginine (a) following a single oral dose and (b) following administration of multiple oral doses of L-homoarginine.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | 1 Month
  To determine the Cmax of L-homoarginine (a) following a single oral dose and (b) following administration of multiple oral doses of L-homoarginine.
Half life of plasma concentration (t1/2) | 1 Month
  To determine the t1/2 of L-homoarginine (a) following a single oral dose and (b) following administration of multiple oral doses of L-homoarginine.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer H Böger, Prof. Dr., Principal Investigator — UHHamburg Eppendorf

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atzler D, Schwedhelm E, Choe CU. L-homoarginine and cardiovascular disease. Curr Opin Clin Nutr Metab Care. 2015 Jan;18(1):83-8. doi: 10.1097/MCO.0000000000000123. PMID 25474016
- [Background] Atzler D, Schonhoff M, Cordts K, Ortland I, Hoppe J, Hummel FC, Gerloff C, Jaehde U, Jagodzinski A, Boger RH, Choe CU, Schwedhelm E. Oral supplementation with L-homoarginine in young volunteers. Br J Clin Pharmacol. 2016 Dec;82(6):1477-1485. doi: 10.1111/bcp.13068. Epub 2016 Sep 20. PMID 27434056